CLINICAL TRIAL: NCT00969423
Title: Chronic Pain After VATS Surgery for Pneumothorax
Brief Title: Chronic Pain After Video-assisted Thoracoscopic Surgery (VATS) Surgery for Pneumothorax
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Rigshospitalet, Denmark, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-A-2009-054
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Pneumothorax
Keywords: persistent pain; neuropathic pain; Chronic Pain; VATS; Primary spontaneous pneumothorax patients
MeSH Terms: conditions — Pneumothorax; Neuralgia; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5 mm equipment (Experimental): 5 mm videoscopic equipment
  Interventions: Device: 5mm videoscope
- 10 mm (Experimental): Use of standard 10 mm VATS equipment
  Interventions: Device: 10mm videoscope

INTERVENTIONS:
Device: 5mm videoscope — use of 5mm videoscope
  Arms: 5 mm equipment
Device: 10mm videoscope — use of 10mm videoscope
  Arms: 10 mm

SUMMARY:
The study will investigate characteristics of chronic pain after VATS surgery with two different sizes of videoscopic equipment.

ELIGIBILITY:
Inclusion Criteria:

* PSP
* Able to understand and give consent
* Can read
* Residing in Denmark

Exclusion Criteria:

* Unable to understand the written information in Danish
* Abuse (Medicine, Drugs, Alcohol)
* Severe psychiatric Illness
* Conflicting neurological disease
* Conversion to open surgery
* Use of neuroaxial analgesia
* Use of electric cauterizer necessitated
* Additional thoracic surgery in the investigation period

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
QST score | 2 years
Post surgical pain | 2 years

SECONDARY OUTCOMES:
Patient related factors, depression, coping etc. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kim Wildgaard, MD, Principal Investigator — Section for Surgical Pathophysiology 4074 Copenhagen, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Wildgaard K, Ravn J, Kehlet H. Chronic post-thoracotomy pain: a critical review of pathogenic mechanisms and strategies for prevention. Eur J Cardiothorac Surg. 2009 Jul;36(1):170-80. doi: 10.1016/j.ejcts.2009.02.005. PMID 19307137